CLINICAL TRIAL: NCT02860754
Title: The Prognostic Capabilities Of A Preoperative Six-Minute Walk Test To Independently Inform Cardiovascular Risk After Major Noncardiac Surgery: Prospective Cohort Study
Brief Title: The Prognostic Capabilities Of A Preoperative Six-Minute Walk Test To Independently Inform Cardiovascular Risk After Major Noncardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Amal Bessissow, MD, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5392
Record Dates: First submitted 2016-04-14; First posted 2016-08-09 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Noncardiac Surgery; Postoperative Myocardial Infarction; Postoperative Death; Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Six-minute walk test (Other): All patients will perform six-minute walk test before surgery, in the preoperative clinic
  Interventions: Other: Six-minute walk test to perform before surgery

INTERVENTIONS:
Other: Six-minute walk test to perform before surgery — During the outpatient preoperative assessment, eligible patients will perform the six-minute walk test.

SUMMARY:
This prospective cohort study aims to determine whether the addition of the 6MWT to the RCRI score improves the risk prediction of postoperative cardiovascular outcomes after noncardiac surgery. In addition, this study will assess whether the patients' reported MET score corresponds to the determined MET score from the 6MWT distance completed.

DETAILED DESCRIPTION:
Study investigators propose to undertake a prospective cohort study at the preoperative clinics of the Royal-Victoria and Montreal General Hospitals of McGill University Health Centre. All patients with planned noncardiac surgery under general or regional anesthesia will be considered for inclusion.

Eligible consenting patients will undergo the 6MWT during their preoperative clinical visit, typically occurring within a few weeks before surgery. This test will be performed by a trained health care worker. Patients will walk back and forth along a 20 m corridor, while attempting to cover as much ground as possible in 6 minutes. Patients will be allowed to rest on the chairs while performing the test if necessary. Patients will be encouraged to resume walking as soon as patients feel physically able. The total covered distance in 6 minutes will be measured to the nearest meter.

The RCRI score will be calculated for each study participant.

ELIGIBILITY:
Inclusion Criteria:

All patients fulfilling all the following inclusion criteria will be enrolled:

* Patients aged ≥ 50 year old and undergoing elective noncardiac surgery, under general anesthesia or regional anesthesia.
* Patients with planned surgery within 3 months of the preoperative visit.

Patients with at least one of the following medical conditions:

* Hypertension, diabetes mellitus, dyslipidemia, coronary artery disease, chronic kidney disease, transient ischemic attack, stroke, or peripheral vascular disease.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

* Patients with a condition preventing mobilization for 6 minutes.
* Patients with significant cardiac disease (e.g., low-threshold angina (angina that occurs with minimal exertion), severe aortic stenosis).
* Patients with severe pulmonary disease restricting mobility.
* Patients refusing to participate.
* Patients previously enrolled in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Measure the additive prognostic value of 6MWT to the RCRI score | At 30 day after surgery
  Investigate the additive prognostic value of the 6MWT to the RCRI score for predicting major cardiovascular complications at 30 day after surgery, in patients undergoing noncardiac surgery.

SECONDARY OUTCOMES:
Compare self reported MET score to 6MWT distance | At preoperative clinic visit. Only one measure
  Determine whether the MET score reported by the patient is comparable to the MET score derived from the 6MWT distance covered.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Bessissow, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada